CLINICAL TRIAL: NCT00691041
Title: A Network Intervention for Reducing Sexual Risk for HIV With African American Men Who Have Sex With Men (AA MSM)
Acronym: UDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-5221
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: HIV Prevention; Men who have sex with men; African American; Unprotected sex; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality; Unsafe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HIV/STI counseling and testing and a 7 session intervention to increase participants' level of knowledge and skills concerning HIV prevention (to decrease HIV acquisition or transmission) and to diffuse the information to their social network
  Interventions: Behavioral: Unity in Diversity
- 2 (No Intervention): HIV/STI counseling and testing and a single 15 minute session of resources available in the community

INTERVENTIONS:
Behavioral: Unity in Diversity — HIV/STI counseling and testing and a 7 session intervention to increase participants' level of knowledge and skills concerning HIV prevention (to decrease HIV acquisition or transmission) and to diffuse the information to their social network
  Arms: 1

SUMMARY:
The purpose of the study is to examine the efficacy of a network-oriented "outreach intervention" to reduce HIV and sexually transmitted infection (STI) related risk behaviors among African American men who have sex with men (AA MSM)and their social network. The hypothesis is to determine whether the new intervention is more efficacious at reducing high risk sexual behaviors than the standard normal of care provided to the public (a single session of individual HIV counseling and testing.

DETAILED DESCRIPTION:
The intervention increases participants' personal level of knowledge and skills concerning HIV prevention and inspires participants to diffuse the information to their social network.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a black / African American male
* Report sex with at least 2 people in past 3 months/ 1 being male
* Willingness to take HIV test or provide documentation if HIV+
* Willingness to identify and recruit friend/relative to study

Exclusion Criteria:

* Under age 18
* Identify as female or transgender
* Not identify as Black / African American

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To increase participants knowledge of HIV/STI risks to assist with decreasing high risk sex/drug behaviors | 3 months after completing intervention

SECONDARY OUTCOMES:
To increase participants' level of knowledge and skills concerning HIV/STI prevention and diffusing the information to their social network) | 3 months after completing the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, PhD, Principal Investigator — Johns Hopkins University -Bloomberg School of Public Health
Locations (1):
- Lighthouse, Baltimore, Maryland, United States

REFERENCES:
- [Result] Tobin KE, German D, Spikes P, Patterson J, Latkin C. A comparison of the social and sexual networks of crack-using and non-crack using African American men who have sex with men. J Urban Health. 2011 Dec;88(6):1052-62. doi: 10.1007/s11524-011-9611-4. PMID 21882072
- [Result] Latkin C, Yang C, Tobin K, Penniman T, Patterson J, Spikes P. Differences in the social networks of African American men who have sex with men only and those who have sex with men and women. Am J Public Health. 2011 Oct;101(10):e18-23. doi: 10.2105/AJPH.2011.300281. Epub 2011 Aug 18. PMID 21852650
- [Result] Latkin C, Yang C, Tobin K, Roebuck G, Spikes P, Patterson J. Social network predictors of disclosure of MSM behavior and HIV-positive serostatus among African American MSM in Baltimore, Maryland. AIDS Behav. 2012 Apr;16(3):535-42. doi: 10.1007/s10461-011-0014-z. PMID 21811844